CLINICAL TRIAL: NCT02187757
Title: A Prospective, Double Blind, Placebo-Controlled, Randomized, Multicentric, Study to Evaluate the Safety, Efficacy and Tolerability of PreLipid®, a Twice-daily Nutritional Supplement in Subjects With Higher Than Normal Blood Lipid Levels
Brief Title: Study to Evaluate Efficacy and Safety of PreLipid® on Subjects With Higher Than Normal Blood Lipid Levels
Acronym: Prelip
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PreEmptive Meds, Pvt. Ltd (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Joe Fenn, Chairman, Department of Clinical & Preventive Cardiology, Medanta, The Medicity, India
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Prelip/Nutra001/PMI13
Record Dates: First submitted 2014-06-30; First posted 2014-07-11 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Hyperlipidemia
Keywords: Dyslipidemia; High cholesterol; High LDL; Triglycerides
MeSH Terms: conditions — Hyperlipidemias; Dyslipidemias; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PreLipid (Experimental): Study Dietary Supplement (PreLipid 600 mg capsules) will be given to subjects twice daily 30 mins before food for 90days along with lifestyle modification.
  Interventions: Dietary Supplement: Study Dietary Supplement (Prelipid 500 mg capsules)
- Placebo 600 mg capsules (Placebo Comparator): Placebo was given to patients twice daily 30 mins before food for 90 days along with lifestyle modification program.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Study Dietary Supplement (Prelipid 500 mg capsules) — Study Dietary Supplement (PreLipid 600 mg capsules) will be given to subjects twice daily 30 mins before food for 90 days along with lifestyle modification.
  Other Names: PreLipid, Natural Cholesterol Supplement, Predisease
  Arms: PreLipid
Dietary Supplement: Placebo
  Other Names: Placebo 600 mg capsules
  Arms: Placebo 600 mg capsules

SUMMARY:
Study to evaluate Efficacy and Safety of PreLipid® on subjects with higher than normal blood lipid levels

DETAILED DESCRIPTION:
A Prospective, Double Blind, Placebo-Controlled, Randomized, Multicentric, study to evaluate the safety, efficacy and tolerability of PreLipid®, a twice-daily nutritional supplement in subjects with higher than normal blood lipid levels

ELIGIBILITY:
Inclusion Criteria:

Newly diagnosed Male or Female participants with higher than normal cholesterol levels defined by the American Heart Association, National Cholesterol Education Program (NCEP) and ATP-III goals for LDL cholesterol and cut off points for therapeutic lifestyle changes (TLCs) and drug therapy in different risk categories:

1. Age ≥ 18 years to ≤ 65 years
2. LDL cholesterol levels >120mg/dl
3. Ability to understand and willingness to sign and date a written Informed Consent Document at the screening visit before any protocol- specific procedures are performed and willing to adhere to the protocol and entire trial procedures -

Exclusion Criteria:

1. Stroke, myocardial infarction, coronary artery bypass graft (CABG) percutaneous transluminal coronary angioplasty (PTCA) or angina pectoris in the past.
2. Cardiac status New York Heart Association class III-IV
3. Uncotrolled blood pressure > 150 mmhg systolic and > 100 mmhg diastolic
4. Impaired renal function as shown by but not limited to serum creatinine ≥ 1.5 mg/dl for males and ≥ 1.4 mg/dl for female
5. Clinically significant peripheral edema
6. Clinical evidence of active liver disease or serum alenine aminotransferase (ALT) or aspartate amino transferase (AST) 2.5 times the upper limit of the normal range (2.5 X ULN)
7. Participants on steroid
8. Pregnancy or lactating women
9. Known hypersensitivity to any of the study drugs
10. Any malignancy within the last 5 years, with exception of adequately treated basal or squamous cell carcinoma of the skin or adequately treated carcinoma insitu.
11. Current addiction or current alcohol abuse or history of substance or alcohol abuse within the last 2 years
12. Subject is the investigator or any sub-investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol
13. Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study.
14. Subject unlikely to comply with protocol e.g. uncooperative attitude, inability to return for follow up visits and unlikelihood completing of the study
15. Any disease or condition that in the opinion of the investigator and/or sponsor may interfere with the completion of the studyevaluation.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of Dietary Supplement PreLipid 600 mg twice-daily in lowering LDL-C levels | Day 1 (Baseline) to Day 90 (End of Study)
  Change in LDL-C % from baseline (Day 1) to the end of supplementation/treatment after 90 days
Safety of Dietary Supplement PreLipid 600 mg twice-daily | Day 1(Baseline) to Day 90 (End of Study)
  Measure changes in Liver Function Tests: Aspartate Aminotransferase (AST) from baseline (Day 1) to End of Study (Day 90); Alanine Aminotransferase (ALT) from baseline (Day 1) to End of Study (Day 90) and Alkaline Phosphatase (ALP) from baseline (Day 1) to End of Study (Day 90)

SECONDARY OUTCOMES:
Changes in Glycemic Status | Day 1 (Baseline) to Day 90 (End of Study)
  To assess percentage changes in Blood Sugar profile (HbA1c) from baseline to at the end of supplementation after 03 months.

OTHER OUTCOMES:
Safety of Dietary Supplement PreLipid 600 mg twice-daily with Kidney Function | Baseline (Day 1) to End of Study (Day 90)
  Measure changes in Renal Function Tests: Blood Urea Nitrogen (BUN) from baseline (Day 1) to End of Study (Day 90); Serum Creatinine from baseline (Day 1) to End of Study (Day 90)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Kasliwal, MD, DM, FIMSA, Study Chair — Medanta, The Medicity, India
Locations (8):
- India (8):
  - Life Care Institute of Medical Science & Research, Ahmedabad, Gujarat
  - Bhatia Hospital Medical Research Society, Mumbai, Maharashtra
  - Dr. Vikas Govind Pai Clinical Research Foundation, Pune, Maharashtra
  - Division of Clinical & Preventive Cardiology, Heart Institute, Gurgaon, National Capital Territory of Delhi
  - Fortis Escorts Hospital, Jaipur, Rajasthan
  - Pace Clinical Research Center, Bangalore, Tamil Nadu
  - Singvi Health Centre, Chennai, Tamil Nadu
  - Rangammal Hospital, Tiruvannamalai, Tamil Nadu